CLINICAL TRIAL: NCT03907007
Title: Effect of Auricular Stimulation on Locomotion in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inventram (Industry)
Collaborators: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Par-03
Record Dates: First submitted 2019-03-29; First posted 2019-04-08 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: Neurostimulator
MeSH Terms: conditions — Parkinson Disease | interventions — Transcutaneous Electric Nerve Stimulation; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sole Medication (No Intervention): Monitoring under current prescribed medication
- Combined stimulation & medication (Active Comparator): Concurrent usage of stimulation with the prescribed medication
  Interventions: Device: Percutaneous electrical nerve stimulation
- Sole Stimulation (Active Comparator): Alternating usage of stimulation to the prescribed medication
  Interventions: Device: Percutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Percutaneous electrical nerve stimulation — Stimulation and medication at the same instant
  Other Names: Stimulation & Medication
  Arms: Combined stimulation & medication
Device: Percutaneous electrical nerve stimulation — Stimulation is given without administering medication
  Other Names: Stimulation Only
  Arms: Sole Stimulation

SUMMARY:
The effect of auricular stimulation on the locomotion capability in patients with Parkinson's Disease was investigated.

DETAILED DESCRIPTION:
Effect of the auricular stimulation as a supplementary and alternative usage to Levodopa was investigated in this study. Clinical data were collected through motion capture system while the participants performed the clinical task asked by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* H&Y Stage >= 1
* Existing bradykinesia symptoms
* Existence of one of the symptoms below
* Resting Tremor
* Rigidity
* Walking disorder

Exclusion Criteria:

* Cardiac Pacemaker
* Psychiatric diagnosis
* Irregular heart/respiration rate
* Pregnancy
* Alcohol consumption
* Cardiovascular disease history
* Wearing an electro-active prosthesis
* Brain surgery history
* Ongoing TENS/PENS therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Stride length [m] | Time Frame: Baseline
  Measurement through motion capture system
Stride length [m] | Time Frame: 20 minutes after stimulation is initiated
  Measurement through motion capture system
Stride length [m] | Time Frame: 40 minutes after stimulation is initiated
  Measurement through motion capture system
Stride length [m] | Time Frame: 60 minutes after stimulation is initiated
  Measurement through motion capture system
Stride velocity [m/s] | Time Frame: Baseline
  Measurement through motion capture system
Stride velocity [m/s] | Time Frame: 20 minutes after stimulation is initiated
  Measurement through motion capture system
Stride velocity [m/s] | Time Frame: 40 minutes after stimulation is initiated
  Measurement through motion capture system
Stride velocity [m/s] | Time Frame: 60 minutes after stimulation is initiated
  Measurement through motion capture system
Turning Velocity [deg/s] | Time Frame: Baseline
  Measurement through motion capture system
Turning Velocity [deg/s] | Time Frame: 20 minutes after stimulation is initiated
  Measurement through motion capture system
Turning Velocity [deg/s] | Time Frame: 40 minutes after stimulation is initiated
  Measurement through motion capture system
Turning Velocity [deg/s] | Time Frame: 60 minutes after stimulation is initiated
  Measurement through motion capture system
Double Support Percentage during walking [%] | Time Frame: Baseline, 20 minutes, 40 minutes, 60 minutes
  Measurement through motion capture system
Double Support Percentage during walking [%] | Time Frame: 20 minutes after stimulation is initiated
  Measurement through motion capture system
Double Support Percentage during walking [%] | Time Frame: 40 minutes after stimulation is initiated
  Measurement through motion capture system
Double Support Percentage during walking [%] | Time Frame: 60 minutes after stimulation is initiated
  Measurement through motion capture system
Swing Phase Percentage during walking [%] | Time Frame: Baseline
  Measurement through motion capture system
Swing Phase Percentage during walking [%] | Time Frame: 20 minutes after stimulation is initiated
  Measurement through motion capture system
Swing Phase Percentage during walking [%] | Time Frame: 40 minutes after stimulation is initiated
  Measurement through motion capture system
Swing Phase Percentage during walking [%] | Time Frame: 60 minutes after stimulation is initiated
  Measurement through motion capture system
Stance Phase Percentage during walking [%] | Time Frame: Baseline, 20 minutes, 40 minutes, 60 minutes
  Measurement through motion capture system
Stance Phase Percentage during walking [%] | Time Frame: 20 minutes after stimulation is initiated
  Measurement through motion capture system
Stance Phase Percentage during walking [%] | Time Frame: 40 minutes after stimulation is initiated
  Measurement through motion capture system
Stance Phase Percentage during walking [%] | Time Frame: 60 minutes after stimulation is initiated
  Measurement through motion capture system

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf O Cakmak, MD, PhD, Principal Investigator — Otago University
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cakmak YO, Ozsoy B, Ertan S, Cakmak OO, Kiziltan G, Yapici-Eser H, Ozyaprak E, Olcer S, Urey H, Gursoy-Ozdemir Y. Intrinsic Auricular Muscle Zone Stimulation Improves Walking Parameters of Parkinson's Patients Faster Than Levodopa in the Motion Capture Analysis: A Pilot Study. Front Neurol. 2020 Oct 7;11:546123. doi: 10.3389/fneur.2020.546123. eCollection 2020. PMID 33117256